CLINICAL TRIAL: NCT00570479
Title: Prevention of Steroid-induced Glaucoma Using Anecortave Acetate
Brief Title: Prophylactic Anecortave Acetate in Patients With a Retisert Implant
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Texas Retina Associates (Other)
Collaborators: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Texas Retina DC-02
Record Dates: First submitted 2007-12-09; First posted 2007-12-11 (Estimated); Last update posted 2012-06-05 (Estimated); Status verified 2012-06

CONDITIONS: Uveitis, Posterior; Glaucoma
Keywords: Retisert; Uveitis; glaucoma
MeSH Terms: conditions — Uveitis, Posterior; Glaucoma; Uveitis | interventions — anecortave acetate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Active Comparator): 50 mgs of anecortave acetate (0.5 ml of a 10% suspension)
  Interventions: Drug: anecortave acetate
- 2 (Active Comparator): Patients will receive 30 mgs of anecortave acetate (0.5 ml of a 6% suspension)
  Interventions: Drug: anecortave acetate
- 3 (Active Comparator): Patients will receive 24 mgs of anecortave acetate (0.4 ml of a 6% suspension)
  Interventions: Drug: anecortave acetate
- 4 (Active Comparator): Patients will receive 12 mgs of anecortave acetate (0.2 ml of a 6% suspension)
  Interventions: Drug: anecortave acetate

INTERVENTIONS:
Drug: anecortave acetate — Patients will receive the specified dose of anecortave acetate every 4 months in an anterior juxtascleral depot injection

SUMMARY:
Retisert implant is an effective therapy for controlling inflammation in patients with non-infectious posterior uveitis. One of the major complications of this device is the development of elevated intraocular pressure (IOP) following implantation in 60% of patients. Glaucoma filtering is required in over 30% of patients at 2 years. Anecortave acetate (AA) has been shown to reduce steroid induced elevated IOP. The purpose of this study was to evaluate the ability of prophylactic anterior juxtascleral depot administration of AA to prevent this Retisert induced elevated IOP.

DETAILED DESCRIPTION:
Test Article: Anecortave Acetate: 6% and 10% Sterile Suspension

Drug Study Dosage: Patients will receive an injection (0.5 mL, 0.4 mL, or 0.2 mL of the 6% Anecortave Acetate suspension or 0.5 mL of the 10% suspension) of study medication every 4 months.

Active Ingredients: Anecortave Acetate (AL-3789)

Route of Administration: Sub-Tenon injection

Objective(s): To evaluate the safety and efficacy of four dosages (50 mg, 30 mg, 24 mg, or 12 mg) of Anecortave Acetate (AA) for the prevention of steroid-induced intraocular pressure (IOP) elevations caused by Retisert.

Study Population: Approximately 24 patients

Structure: Parallel Group Duration of Treatment: 3 years

Description: Observer-masked study of the safety and efficacy of Anecortave Acetate 6% or 10 % administered by a sub-Tenon injection. Up to 24 patients with recent implantation of a Retisert implant will be given a sub-Tenon injection of either 0.5 mL, 0.4 mL, or 0.2 mL of 6% Anecortave Acetate Sterile suspension or 0.5 mL of the 10% suspension. Patients will receive periodic evaluations and re-treatment every 4 months for as long as 3 years. The end point will be an IOP which requires surgical intervention. An initial assessment of efficacy will be made at 18 months. If any patient treated with a lower dose develops an IOP of greater than 30mHg, then they are eligible to receive the 50 mg dose.

Multicenter: Yes Number of Centers: 1 Masking: Observer masked (IOP-reader)

Method of Patient Assignment:

Randomization: Yes

ELIGIBILITY:
Inclusion Criteria:

Approximately 24 patients with recent implantation of the Retisert implant who meet the inclusion/exclusion criteria defined below will be enrolled in the study. They will be identified from the current and future patients of the clinical practices.

* Patients must be willing to sign an informed consent form, able to make the required study visits, and able to follow instructions.
* Patient must be at least 12 years of age.
* Implantation of a Retisert implant in the last 12 weeks.

Exclusion Criteria:

* Patient has history of any medical condition which would preclude scheduled study visits or completion of the study (i.e., unstable cardiovascular disease)
* Patient has insertion of a scleral buckle in the study eye.
* Patient has known medical history of allergy or sensitivity to the steroid family of drugs.
* Patient is on anticoagulant therapy, with the exception of aspirin and antiplatelet therapy. Patient has a medical history of a bleeding disorder.
* Patient has clinical evidence of scleral thinning.

Ages: 10 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2006-09; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Percentage of patients requiring glaucoma filtering surgery | 3 years

SECONDARY OUTCOMES:
Percentage of patients requiring topical glaucoma medication | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: David G Callanan, MD, Principal Investigator — Texas Retina Associates
Locations (1):
- Texas Retina Associates, Arlington, Texas, United States